CLINICAL TRIAL: NCT07060521
Title: Soft Tissue Mobilization is More Effective Than Self-stretching in Reducing Common Wrist Extensor Tendon Stiffness in Recreational Tennis Players
Brief Title: Differences in Elbow Stiffness Comparing Massage to Stretching in Tennis Players
Acronym: DESMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dayton (Other)
Responsible Party: Principal Investigator, Joseph Day, Associate Professor of Physical Therapy, University of Dayton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20597767
Record Dates: First submitted 2025-06-09; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Tendon Stiffness; Lateral Elbow Tendinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self stretching (Active Comparator)
  Interventions: Other: Self Stretching
- Soft Tissue Mobilization (Experimental)
  Interventions: Other: soft tissue mobilization

INTERVENTIONS:
Other: soft tissue mobilization — massage
  Other Names: self stretching
  Arms: Soft Tissue Mobilization
Other: Self Stretching — self stretching
  Arms: Self stretching

SUMMARY:
Background and Purpose: Shear wave elastography (SWE) provides quantifiable and specific data regarding muscle and tendon stiffness. Increased muscle and tendon stiffness plays a role in the development of musculoskeletal pathologies. A number of interventions have been proposed to temporarily reduce muscle/tendon stiffness including soft tissue mobilization (massage) and stretching.

Purpose: To investigate the effects of soft tissue mobilization versus stretching on tissue stiffness in a group of competitive tennis players.

Participants: Healthy competitive tennis players who meet the inclusion criteria and consent to participate will be assessed and treated at the University of Dayton Department of Physical Therapy.

Methods: All participants will be examined with shear wave elastography to determine the stiffness of the dominant common extensor tendon with the participant in sitting, arm supported and relaxed. A second stiffness measure will be taken 5 minutes after the first measure to determine intra-rater reliability. Participants will be divided into 1 of 2 treatment groups (soft tissue massage or passive stretching) for approximately 5 minutes. Shear wave stiffness measures will be taken immediately after intervention for both groups. Shear wave elastography will be measured one final time following a 15-minute rest period after the intervention

DETAILED DESCRIPTION:
Background:

Soft tissue stiffness, caused by overuse, can lead to movement impairments and is thought to be a causal factor in tennis players developing lateral elbow tendinopathy (LET). The role of eccentric fatigue in activities can be linked to certain overuse conditions. A recent study explored the effect of eccentric fatigue on stretch-shortening cycle effectiveness. The findings of the study indicate that fatigue alters the stretch-shortening cycle. It was found that eccentric fatigue results in an increase in lower limb stiffness along with a decrease in stretch amplitude1. An increase in fatigue can lead to an increased passive load to a tissue, leading to overuse conditions such as LET.

Clinically, tissue stiffness may be assessed with range of motion measures and end feels. However, these techniques are not specific and are difficult to objectify. Shear Wave Elastography (SWE) allows the assessment of tissue stiffness, is non-invasive, and provides quantifiable data3.Through the use of the SWE, tissue elasticity can be measured allowing the ability to test and compare more specific rehabilitation strategies in a static or dynamic setting. SWE is a reliable and diagnostic tool that is sensitive enough to compare the effects of rehabilitation techniques on the mechanical properties of muscle.

There are many techniques used in the conservative management of muscle and tendon stiffness. Perhaps the most common method for decreasing muscle stiffness is manual massage. Soft tissue massage increases blood flow, reduces muscle tension as well as neurological excitability. Soft tissue massage uses mechanical pressure, which in turn will decrease active and passive stiffness within the muscle. For example, a mixture of isometric contraction and instrument-assisted soft tissue mobilization have been shown to also alleviate shoulder stiffness. Instrument-assisted soft tissue massage has also been shown to be effective in regards to improving shoulder horizontal adduction and internal rotation. Other studies have investigated the effectiveness of manual therapy and stretching on muscle and tendon stiffness.8 Therefore both massage and stretching techniques have shown to reduce muscle and tendon stiffness.

A survey of the literature finds few studies that have used SWE technology in evaluation of the efficacy of manual therapies or stretching regimen. Studies that used SWE and included manual therapy did not compare to other interventions and were focused on the lower extremity or the jaw. Research is needed to determine the most effective and efficient technique to promote a decrease in stiffness so that movement impairments and pathology can be avoided. Therefore, the purpose of our study is to will explore the effect of massage and stretching on common wrist extensor tendon stiffness in healthy competitive tennis players.

Methods:

All participants will be examined with shear wave elastography to determine the stiffness of the specified passive structures. The common wrist extensors will be examined on the dominant test side using SWE with the arm in the following resting position: shoulder at 70 degrees of abduction, elbow at 90 degrees of flexion, and forearm in pronation. Three measurements will be taken in this position and the average value will be recorded. Following these measurements, the participant will be given a 5-minute rest. For the purpose of establishing intra-rater reliability, another set of three more measurements using the SWE on the wrist extensor tendon will be taken. After these two initial collections are taken, participants will be randomized to either common wrist extensor stretching or soft tissue massage.

Participants undergoing stretching will be placed in the following position: shoulder at 90 degrees of flexion on plinth, elbow at 0 degrees of extension, and forearm in pronation. Wrist comfort level will be of strong but tolerable stretch length. Participants will be asked to report the comfort level of wrist flexion as tolerable ',' strong but tolerable, 'uncomfortable', or 'intolerable'. The intensity will be maintained at a 'strong but tolerable' level for consistency and efficacy."8 Participants will undergo a self-stretch holding this position for 30 seconds and repeating 5 times. Tendon stiffness will be measured again using SWE in a resting position (shoulder at 70 degrees of abduction, elbow at 90 degrees of flexion, and forearm in pronation). Three measurements will again be taken and the average tissue stiffness measured will be recorded. Participants will then have a 15-minute rest period after the post-intervention measurements. Similar to first three SWE collections, the average of the three measurements will be recorded as the value for this participant.

Participants undergoing deep tissue massage will remain in resting position (shoulder at 70 degrees abducted, elbow 90-degree flexion, and forearm in pronation). Massage will last for 5 minutes consisting of petrissage (a deep kneading) with linked effleurage (more superficial strokes) on the dominant test side. Massage will use a moisturizer (cream, or oil, etc) to minimize patient discomfort from skin friction. Participants will be asked to report the comfort level of the massage as 'completely tolerable', 'strong but tolerable', 'uncomfortable', or 'intolerable'. The intensity will be maintained at a 'strong but tolerable' level for consistency and efficacy."8 After the massage intervention tissue stiffness will be measured again using SWE in the resting position (shoulder at 70 degrees of abduction, elbow at 90 degrees of flexion, and forearm in pronation). Three measurements will again be taken and the average tissue stiffness measured will be recorded. Participants will then have a 15-minute rest period after the intervention measurements. Like the first three collections, the average of the three measurements will be recorded as the value for this participant.

ELIGIBILITY:
Inclusion Criteria:

1. An adult18 - 80 years old.
2. Demonstrate sufficient fluency in spoken or written English to communicate with the research examiner and complete questionnaires.
3. Tennis player at any level playing at least 1 time a week on average

Exclusion Criteria:

1. Prior upper extremity surgery within 6 months of the study's start date
2. Any diagnosed upper extremity pathologies or injuries within 6 months of the study's start date.
3. Rehabilitative/medical treatment of the upper extremity in the past year
4. Unable to tolerate soft tissue massage or stretching treatments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
Tendon Stiffness: 2D shear wave elastography (SWE ultrasound imaging GE Logiq S8, 9L linear transducer) | From enrollment until the end of a single session which is approximately 45 minutes per participant
  Data collection for tendon stiffness will require the use of the following instrument: 2D shear wave elastography (SWE) ultrasound imaging (GE Logiq S8, 9L linear transducer). SWE is a new ultrasound imaging setting that simply determines the hardness or stiffness of a muscle. Ultrasound waves are transmitted through a linear probe to the gel medium and on to the contact surface of the body. SWE is an a measure of the speed at which the ultrasound waves pass through the body. The more dense the material (stiffer), the faster the wave will propagate. The side of the probe indicator along the transducer will be placed directly over the lateral epicondyle while the distal end of the transducer was in line with the middle of the radiocarpal joint. Three images will be taken and stiffness values will be recorded for each image. The shear wave modulus will then be automatically generated in kilopascals (kPa)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Dayton, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
I plan to consider this possibility when submitting a manuscript

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-07-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT07060521/Prot_SAP_000.pdf